CLINICAL TRIAL: NCT05838859
Title: Mental Health and Contraception- Are we Doing Enough? A Study Exploring the Current Practice of Providing Contraceptive Advice by Mental Health Professionals and Service User Experience
Brief Title: Contraception and Mental Health: Are we Doing Enough?
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Surrey and Borders Partnership NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS 284443
Record Dates: First submitted 2022-06-01; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Mental Health Issue; Woman's Health; Contraception; Family Planning

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Female service users of childbearing age: Contraception Advice Experiences Survey - using a self-report questionnaire of female service users.
- Mental health care professionals: Contraception in Mental Health Survey - self-report questionnaire of professionals' current practices, attitude and knowledge

SUMMARY:
The study seeks to determine current practices and perspectives of contraceptive advice of both service users and professionals. It aims to examine 1) the experiences of female service users of reproductive potential with mental health conditions of contraceptive advice from mental health professionals and 2) the current practice of providing contraceptive advice by mental health professionals.

DETAILED DESCRIPTION:
The WHO Sustainable development goals (SDGs) outline the necessity to ensure universal access to sexual and reproductive healthcare services, including family planning information and education, and the integration of reproductive health into national strategies and programmes. Family planning and contraception knowledge is integral to maintaining or improving relationships for well-being. Whilst contraceptive knowledge is undoubtedly important for all reproductive-aged people, it is of increased importance for women with mental health conditions who are considered a "doubly disadvantaged" group due to their gender and diagnosis.

Women can experience significant reproductive health problems including reduced fertility due to pharmacology use, high rates of unplanned pregnancies, safeguarding processes and increased rate of malformations in their offspring.

NICE (National Institute for Health and Care Excellence) guidelines recommend discussing with women of childbearing potential who have or had mental health problems the use of contraception and any plans of pregnancy, how pregnancy and childbirth might affect a mental health problem and how mental health problem and its treatment might affect the women, the foetus or baby. Although international and national legislation clearly acknowledges equal rights for women with disabilities with regards to family planning, they continue to face challenges in accessing these SRH.

Women who experience severe and persistent mental health issues are more likely to experience unplanned pregnancy, maybe likely to engage in sexual risk taking behaviour and are at a higher risk of sexually transmitted diseases. A recent systematic review estimates that in the UK, at any given time, 9-10% of women will be parents with mental disorder. There are well-established links between parental mental disorder and poor outcomes in children, although not all children are at risk. Throughout the period of foetal development, infancy and toddlerhood the brain of a baby is growing and developing.) These first 1001 days are critical because of optimal brain development and also gives the baby the best possible start in life. People who lack nurture from one or more caring adults in the first 1001 days of their lives achieve less in education and in the world of work; are more likely to behave anti-socially, and are less healthy, physically as well as mentally, than individuals who were given a better start. Furthermore, the harm done to them is likely to be perpetuated in an inter-generational cycle when they have children of their own .

The investigators also looked at some more scientific evidence from the point of view of mental health professionals. Mental health professionals are poor at collecting information regarding the parenting status of their patients and tend not to enquire about children's welfare and needs. In addition, mental health professionals report patients' lack of insight regarding the illness and its impact on children, insufficient knowledge and skills and concerns that discussing parenting and child-related issues might impair the relationship they have with their patient. A research study has found that 16% of childbearing age women were prescribed teratogens. For women with mental health conditions who want to avoid unintended pregnancy, effective contraceptive use can be an important strategy to maintain and even improve health and wellbeing. Barriers in the provision of appropriate reproductive advice includes difficulties in determining "best interests", feeling ill-equipped to discuss sexual and reproductive health due to perceived boundaries and embarrassment, and ethical challenges.

Study Design An observational quantitative cross-sectional design study will be utilised. The investigators will not intervene in any way but simply record the answers to questionnaire of the study participants. All the measurements for the participants will be obtained at a single point in time, although recruitment may take place across a longer period. This is the most suitable method for this study as it minimises loss to follow up, obtrusiveness and response bias and will allow for future replicability and comparisons across other NHS Trusts.

Participants / Population This will be a two-armed study sampling service user of childbearing age receiving SABP mental health care services and mental health care professionals. The study will seek to recruit patients from inpatient units and community mental health teams from Surrey and Borders Partnership NHS Foundation Trust (SABP) and Mental health care professionals from the Trust.

ELIGIBILITY:
Inclusion Criteria:

Service Users

* Female aged between 18 and 50 years of age.
* Under SABP mental health services
* Diagnosed DSM IV mental health condition.
* Capacity to give informed consent.

Professionals

* Doctors, nursing staff Band 6 or above, non-medical prescribers and care- coordinators.
* Employed by Surrey and Borders Partnership NHS Foundation

Exclusion Criteria:

Service Users

* Service users under specialist services such as eating disorders, perinatal services, substance misuse services.
* Service users under Child and Adolescent Mental Health services and Learning Disability Mental Health Services.
* Lacking capacity to consent.
* Under 18 or over 50 years of age
* Service users detained under the Mental Health Act in the inpatient unit or under community treatment order(CTO) in the community.

Professionals

* Mental health professionals not employed by Surrey & Borders Partnership Foundation NHS Trust
* Mental health professionals not working in Working Age Adult Services.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The service user survey is only for female service users under Surrey and Borders NHS Trust
Study Population: This will be a two-armed study sampling service user of childbearing age receiving SABP mental health care services and mental health care professionals. The study will seek to recruit patients from inpatient units and community mental health teams from Surrey and Borders Partnership NHS Foundation and Mental health care professionals from the Trust.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-02-09 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-02-01 (Estimated)

PRIMARY OUTCOMES:
Service user experience- online survey - designed by investigators | Sep 2022
  To examine if female service users of childbearing age under the care of mental health services are receiving adequate advice on contraception.
Mental health professionals experience - online survey- designed by investigators | Sep 2022
  To examine the knowledge, practices and attitudes of mental health professionals in providing advice regarding contraception.

CONTACTS AND LOCATIONS:
Overall Officials: Josie Jenkinson, MRCPsych, Principal Investigator — Surrey and Borders Partnership NHS Foundation Trust
Locations (1):
- Surrey and Borders NHS Foundation Trust, Leatherhead, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Arain M, Campbell MJ, Cooper CL, Lancaster GA. What is a pilot or feasibility study? A review of current practice and editorial policy. BMC Med Res Methodol. 2010 Jul 16;10:67. doi: 10.1186/1471-2288-10-67. PMID 20637084
- [Result] Gee B, Notley C, Byrne R, Clarke T, Hodgekins J, French P, Fowler D. Young people's experiences of Social Recovery Cognitive Behavioural Therapy and treatment as usual in the PRODIGY trial. Early Interv Psychiatry. 2018 Oct;12(5):879-885. doi: 10.1111/eip.12381. Epub 2016 Sep 7. PMID 27600941
- [Result] Haslegrave M. Ensuring the inclusion of sexual and reproductive health and rights under a sustainable development goal on health in the post-2015 human rights framework for development. Reprod Health Matters. 2013 Nov;21(42):61-73. doi: 10.1016/S0968-8080(13)42742-8. PMID 24315064
- [Result] Henshaw, C & Protti, C (2010) Addressing the sexual and reproductive health needs of women who use mental health services, and Advances in psychiatric treatment Vol 16, 272 - 278.
- [Result] Howard LM, Megnin-Viggars O, Symington I, Pilling S; Guideline Development Group. Antenatal and postnatal mental health: summary of updated NICE guidance. BMJ. 2014 Dec 18;349:g7394. doi: 10.1136/bmj.g7394. No abstract available. PMID 25523903